CLINICAL TRIAL: NCT00916838
Title: Neurocognitive Impact of Hypoglycemia in Type 1 Diabetes
Acronym: HYPO
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 02-1012 -201102446; R01DK064832 (NIH)
Record Dates: First submitted 2009-06-02; First posted 2009-06-10 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Type 1 Diabetes Mellitis
Keywords: Type 1 Diabetes Mellitis; MRI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 1 Diabetes Mellitis: Children with Type 1 Diabetes Mellitis (T1DM) between 4 and 16 were recruited.
- Non diabetic Control: 62 healthy siblings also enrolled in the study between the ages of 4 and 17.

SUMMARY:
125 children with Type 1 Diabetes mellitis (T1DM) between 4 and 16 were recruited and 62 healthy siblings also enrolled in the study.

Children with T1DM and sibling controls ages 4 to 16 were assessed on memory and executive control skills at entry to the study (Test 1) and after two years of close monitoring for blood sugar events (Test 2). Diabetic children have their blood sugar tested directly before and after cognitive testing to ensure their blood sugar is within range during the testing. The 2-year follow-up period involves parents/child reporting any severe diabetic episode and periodically providing the results of the diabetic child's usual blood tests from their glucose monitoring device.

Children 7 and older also underwent high resolution MRI scans.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 - 16 (for MRI, must be 7 or older)

Exclusion Criteria:

* Pregnant or lactating (females 13+)
* Chronic disease other than T1DM, well-controlled asthma, or Hashimoto's thyroiditis. (Exclude for hypothyroidism)
* Other current serious medical illness
* Co-morbid psychiatric illness: such as mania, ADHD, LD, major depression, mental retardation, or psychoactive drug dependence
* Co-morbid neurological illness: stroke, seizure, major loss of consciousness, other brain trauma/surgery, or head injuries (i.e. near drowning), encephalitis, or hydrocephalus, blindness, deafness
* EXCEPT T1DM-related
* Pre-maturity at birth >4 wks early (<36 wk term) w/ sequelae e.g. on respirator at NICU
* Use of psychoactive medications or exposure to neuroleptics (except that exposures of less than 1 month, occurring more than 5 years ago, will be allowed) or pts. w/recent tx w/dopamine depleting agents or stimulants such as Ritalin, Cylert, Adderall
* Contraindication to MRI scan (e.g. claustrophobia, metal implants, foreign bodies) - N/A if < 4 years old
* Full set (top and bottom) orthodontic braces. (Half set braces, fillings, and retainers are OK)

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 125 children with Type 1 Diabetes Mellitus (T1DM) between 4 and 16 were recruited from the Diabetes Clinic at St. Louis Children's Hospital. 62 healthy siblings between 4 and 16 also enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2003-01; Primary Completion 2006-03 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara G Hershey, PhD., Principal Investigator — Washington Univeristy School of Medicine